CLINICAL TRIAL: NCT06893588
Title: Prospective, Open-Label, Multi-Center ProceDural Data CollectIon Case Registry on NeVa VS for CerebraL VAsospasm ManagemenT in Post SAH PatiEnts (The DILATE Registry)
Brief Title: Registry on NeVa VS for CerebraL VAsospasm ManagemenT in Post SAH PatiEnts
Acronym: DILATE
Status: Not yet recruiting | Type: Observational
Sponsor: Vesalio (Industry)
Responsible Party: Sponsor
Other Study IDs: VS-011
Record Dates: First submitted 2025-02-03; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Cerebral Vasospasm; Aneurysmal Subarachnoid Hemorrhage (aSAH)
Keywords: vasospasm
MeSH Terms: conditions — Vasospasm, Intracranial; Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Treatment Group
  Interventions: Device: NEVA VS

INTERVENTIONS:
Device: NEVA VS — cerebral artery dilation device

SUMMARY:
A multi-center, observational registry study intended to assess the HDE-approved NeVa VS cerebral artery dilation device in patients with symptomatic cerebral vasospasm caused by aneurysmal subarachnoid hemorrhage (aSAH)

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥22
2. Symptomatic cerebral vasospasm secondary to aneurysmal subarachnoid hemorrhage (aSAH) in the internal carotid artery (ICA), middle cerebral artery (MCA), anterior cerebral artery (ACA), posterior cerebral artery (PCA), or basilar artery (BA)
3. Vessel dilation procedure was performed with the NeVa VS
4. Subject or legal representative is able and willing to give informed consent within 3 days (72 hours) post-index procedure

Exclusion Criteria:

* None

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects with cerebral vasospasm
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-04-14 (Estimated); Primary Completion 2027-02-14 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Improvement in target vessel diameter following NeVa VS use | Up to 1 hour post procedure

IPD SHARING:
Plan to Share IPD: No